CLINICAL TRIAL: NCT00940290
Title: Different Grading Systems to Grade Evidence and Recommendations in Clinical Practice Guidelines: Does it Influence the Clinicians´ Behavior?
Brief Title: Practice Guidelines Grading Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Responsible Party: Carlos Alberto Cuello-Garcia, Instituto Tecnologico y de Estudios Superiores de Monterrey
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CMBE-ITESM-1
Record Dates: First submitted 2009-07-13; First posted 2009-07-16 (Estimated); Results first posted 2010-01-13 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-11

CONDITIONS: Decision Making
Keywords: practice guideline as topic; decision making; evidence based medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- GRADE system (Other): A clinical recommendation built and graded with the GRADE working group system
  Interventions: Other: Graded Clinical Recommendation
- SIGN grading system (Other): A clinical recommendation built and graded with the Scottish Intercollegiate Guidelines Network system
  Interventions: Other: Graded Clinical Recommendation
- NICE grading system (Other): A clinical recommendation built and graded with National Institute of Clinical Excellence grading system
  Interventions: Other: Graded Clinical Recommendation
- CEBM-Oxford (Other): A clinical recommendation built and graded with the Centre for Evidence-Based Medicine grading system
  Interventions: Other: Graded Clinical Recommendation

INTERVENTIONS:
Other: Graded Clinical Recommendation — Graded recommendation in reference to a clinical condition written as it would be in a clinical practice guideline

SUMMARY:
Clinical practice guidelines (CPG) are systematically developed statements to assist practitioner and patient decisions about appropriate health care for specific clinical circumstances. They are developed to give a recommendation based on the best evidence available. Through a randomized trial, the investigators intend to provide information about which of the four grading systems most used today to grade evidence and recommendations in CPGs, could change physician´s behavior towards a common clinical situation in daily practice.

DETAILED DESCRIPTION:
Clinical practice guidelines (CPG) are used by professional and consumer organizations who are demanding more rigorous processes to ensure that health decisions are well informed by the best available research evidence. More than 60 different grading systems are used today to grade evidence and recommendations in CPGs. The investigators aimed to provide information about which of the four most common grading systems used today (GRADE, SIGN, NICE and CEBM-Oxford) could change physician´s behavior when reading a clinical recommendation in a CPG. The investigators will randomize 216 pediatricians and pediatricians in training into four groups (one for each grading system) to read a clinical case and to make a decision before reading the CPG statement graded with any of the four grading systems. After that they will re-consider their answer and post a new one based on the graded recommendation. The investigators will measure change in their decision and among groups.

ELIGIBILITY:
Inclusion Criteria:

* Pediatricians and residents in pediatrics

Exclusion Criteria:

* Less than six months in clinical practice

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Cuello-Garcia, MD, Principal Investigator — Instituto Tecnologico y de Estudios Superiores de Monterey
Locations (1):
- Escuela de Medicina y Biotecnologia del ITESM, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Derived] Cuello Garcia CA, Pacheco Alvarado KP, Perez Gaxiola G. Grading recommendations in clinical practice guidelines: randomised experimental evaluation of four different systems. Arch Dis Child. 2011 Aug;96(8):723-8. doi: 10.1136/adc.2010.199307. Epub 2011 May 19. PMID 21596725

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric residents, pediatricians and sub-specialists were recruited from their clinical practices to participate in the study. All in known teaching hospitals in Monterrey and Mexico city. Recruitment from September 1st to October 21st.
Pre-assignment Details: Participants were not eligible for randomization if they refuse to participate in the trial or if they reported less than six months of clinical practice (residents). After randomization they were allocated to one of the four study groups. A survey was applied and no wash out was observed or desertions.
Period: Overall Study
Arm/Group | GRADE System | SIGN Grading System | NICE Grading System | CEBM-Oxford
Started | 54 | 53 | 55 | 54
Completed | 54 | 53 | 55 | 54
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GRADE System | SIGN Grading System | NICE Grading System | CEBM-Oxford | Total
Number analyzed (Participants) | 54 | 53 | 55 | 54 | 216
Age Continuous [Median (Inter-Quartile Range); unit: years] | 30 [28 to 47] | 34 [28 to 47] | 31 [28 to 40] | 38 [28 to 49] | 32 [28 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 25 | 25 | 102
  Male | 29 | 26 | 30 | 29 | 114
Years of practice [Median (Inter-Quartile Range); unit: Years]
  Years of practice | 4 [2 to 19] | 5 [2 to 18] | 4 [2 to 12] | 9 [2 to 20] | 5 [2 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Change in Behavior in Physicians Attitude Towards a Decision to Give a Medication
Description: A fictitious clinical case of a child with acute diarrhea was presented. The physician read the case and then answered the question "would you recommend racecadotril to this patient?" A zero to 10 visual-analog scale and a Likert scale were used to measure the decision of the physician related to the clinical case presented (from zero="definitely no" to 10="definitely yes"). Mean differences before-after and among groups were measured on the 10 centimeters scale.
Time Frame: One day
Measure: Mean (95% Confidence Interval); unit: Mean change in centimeters
Arm/Group | GRADE System | SIGN Grading System | NICE Grading System | CEBM-Oxford
Number analyzed (Participants) | 54 | 53 | 55 | 54
Mean change in centimeters | 2.18 [1.48 to 2.88] | 0.31 [-0.41 to 1.05] | 0.04 [-0.68 to 0.77] | 0.08 [-0.52 to 0.69]
Statistical Analysis 1: Comparison: GRADE System vs SIGN Grading System vs NICE Grading System vs CEBM-Oxford; After reading the clinical practice guideline, the median response from the four groups were compared using the Kruskal-Wallis statistic; Test type: Superiority or Other; p = 0.007, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Do not apply
Description: As this is a survey in a randomized group of physicians, we do not expect to see adverse events
Arm/Group | GRADE System | SIGN Grading System | NICE Grading System | CEBM-Oxford
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The outcome was measured in only one topic and could be not expanded to other areas of pediatrics or even other specialties in medicine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes